CLINICAL TRIAL: NCT04073017
Title: Proprietary Amino Acid-Based Medical Food (Enterade) in Carcinoid Syndrome and Non-Carcinoid Syndrome Neuroendocrine Tumor Patients With Quality of Life Limiting Bowel Frequency
Brief Title: Enterade in Carcinoid/Non-Carcinoid Syndrome Neuroendocrine Tumor Patients With Quality of Life Limiting Bowel Frequency
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: Entrinsic Bioscience Inc. (Industry)
Responsible Party: Principal Investigator, Satya Das, Sponsor Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VICC GI 1943
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Neuroendocrine Tumor; Carcinoid Syndrome
MeSH Terms: conditions — Neuroendocrine Tumors; Serotonin Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enterade (Experimental): Carcinoid Syndrome: Participants will drink a bottle of Enterade two time per day for 4 weeks.
  Interventions: Dietary Supplement: Enterade®; Other: Functional Assessment of Chronic Illness Therapy for Patients with Diarrhea (version 4.0)
- Experimental (Experimental): Non-Carcinoid Syndrome: Participants will drink a bottle of Enterade two time per day for 4 weeks.
  Interventions: Dietary Supplement: Enterade®; Other: Functional Assessment of Chronic Illness Therapy for Patients with Diarrhea (version 4.0)

INTERVENTIONS:
Dietary Supplement: Enterade® — Participants will drink an 8 ounce bottle of Enterade® twice a day for 4 weeks
Other: Functional Assessment of Chronic Illness Therapy for Patients with Diarrhea (version 4.0) — Ancillary studies
  Other Names: FACIT-D

SUMMARY:
This is an open-label phase II basket study evaluating the ability of enterade® to reduce bowel frequency in neuroendocrine tumor (NET) patients with carcinoid syndrome and non-carcinoid syndrome.

DETAILED DESCRIPTION:
Primary Objective:

- To assess the ability of enterade to reduce bowel movement frequency in NET patients with and without carcinoid syndrome.

Secondary Objectives:

* To assess subject-reported health-related quality of life measures in subjects before and after compound administration.
* To characterize the side effect profile and tolerability of the compound as measured by the number of total 8-oz enterade® bottles consumed throughout the trial.
* To evaluate changes in serum electrolytes before and after administration of the compound.
* To assess differences in intravenous fluid requirement and/or hospitalizations for dehydration in patients between observation period and active enterade® period.
* To evaluate differences in utilization of standard-of-care anti-diarrheal medications in patients between observation period and enterade® period.
* To compare subjective bloating and flatulence in patients before and after administration of the compound.
* To evaluate changes in patient weight before and after administration of the compound.

Exploratory Objectives:

* To assess changes in serum and stool inflammatory markers before and after the study compound.
* To evaluate changes in fecal lactoferrin before and after study compound administration.

ELIGIBILITY:
Inclusion Criteria:

Carcinoid syndrome:

Participants must have histopathologically confirmed neuroendocrine tumor with 4 or more bowel movements per day on standard anti-diarrheal regimen (which includes somatostatin analogs and/or Telotristat Ethyl). Additionally, a plasma 5-HIAA, or a urine 24-hour 5-HIAA or plasma secretory hormone levels (VIP, gastrin) above the upper limit of normal per reference lab. Patients may be grouped into this cohort based on a previous plasma 5-HIAA level though the final cohort determination will be made based upon the 5-HIAA level drawn during screening.

Non-Carcinoid Syndrome:

Participants who have histopathologically confirmed neuroendocrine tumor and have 4 or more bowel movements per day on standard anti-diarrheal regimen (which may or may not include somatostatin analogs), but do not have elevated results for one of the following: plasma 5-HIAA, or 24-hour urine 5-HIAA or other plasma secretory hormone levels (VIP, gastrin) above the upper limit of normal per reference lab. Patients may be grouped into this cohort based on a previous plasma 5-HIAA level though the final cohort determination will be made based upon the 5-HIAA level drawn during screening

* ECOG performance status ≤ 2 (Karnofsky ≥60%)
* Ability to tolerate thin liquids by mouth at the time of enrollment.
* Ability to understand and the willingness to sign a written informed consent document.
* Subject who are willing to take enterade® as instructed will be eligible.

Exclusion Criteria:

* Known allergy to Stevia.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active
* Clostridium difficile infection or history of Clostridium difficile infection.
* Participants with a history of inflammatory bowel disease, irritable bowel syndrome, bariatric surgery and/or Celiac disease.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* Patients who have had enterade® within the past 3 months.
* Pregnant or breastfeeding women. The safety of enterade® has not been validated in this patient population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
Change in bowel movement frequency | At 8 weeks
  Changes in number of average daily bowel movements from baseline

SECONDARY OUTCOMES:
Health-Related Quality of Life: Functional Assessment of Chronic Illness Therapy for Patients with Diarrhea (FACIT-D) version 4.0 | At 8 weeks
  The FACIT-D is a questionnaire composed of 5 categories (physical well-being, social/family well-being, emotional well-being, functional well-being and additional concerns). Each category has 6-11 questions which are scored on a 0 (not at all) to 4 (very much) scale. Groups of categories are scored differently. For example in the additional concerns, emotional well-being and physical well-being categories, a higher score reflects poorer quality of life. In the family well-being and functional well-being categories, a higher score indicates better outcomes.
Tolerability of enterade®: number of enterade® drinks consumed | At 8 weeks
  Measured by the total number of enterade® drinks consumed
Incidents adverse events | At 8 weeks
  NCI CTCAE version 5.0
Change in serum electrolytes (Sodium) | At 8 weeks
  The electrolyte sodium will be assessed for each patient before and after enterade® (measured in mmol/L)
Change in serum electrolytes (Potassium) | At 8 weeks
  The electrolyte potassium will be assessed for each patient before and after enterade® (measured in mmol/L)
Change in serum electrolytes (Chloride) | At 8 weeks
  The electrolyte chloride will be assessed for each patient before and after enterade® (measured in mmol/L)
Change in serum electrolytes (Magnesium) | At 8 weeks
  The electrolyte magnesium will be assessed for each patient before and after enterade® (measured in mg/dL )
Change in serum electrolytes (Phosphorous) | At 8 weeks
  The electrolyte phosphorous will be assessed for each patient before and after enterade® (measured in mg/dL )
Differences in intravenous fluid requirements | At 8 weeks
  Measured by the number of incidence requiring intravenous fluid before and after taking enterade®
Differences in use of standard-of-care anti-diarrhea medications | At 8 weeks
  Measured by reported incidence of standard-of-care anti-diarrhea medications usage before and after taking enterade®
Differences in bloating | At 8 weeks
  Measured by reported incidence of bloating before and after taking enterade®
Differences in flatulence | At 8 weeks
  Measured by reported incidence of flatulence before and after taking enterade®
Changes in weight | At 8 weeks
  Measured by fluctuation in weight before and after taking enterade®

CONTACTS AND LOCATIONS:
Overall Officials: Satya Das, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No